CLINICAL TRIAL: NCT06428474
Title: Effectiveness of Oral Health Educational Program on the Knowledge and Practice of Institutionalized Orphan Children in Alexandria, Egypt
Brief Title: Implementation of Oral Health Educational Program on Orphan Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Inas Karawia, Lecturer, Faculty of Dentistry, Pharos University, Pharos University in Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UREAC-04-3-219
Record Dates: First submitted 2024-05-09; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Dental Caries; Knowledge; Practice
Keywords: Oral health education; knowledge; practice; oral hygiene
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children who are living in orphanages (Experimental): Orphan children aged 6-12
  Interventions: Other: Health education

INTERVENTIONS:
Other: Health education — Oral health education program designed for orphans children

SUMMARY:
Oral diseases are most prevalent among children. Orphans children are one of the most vulnerable groups to diseases especially oral diseases.

Knowledge toward oral cavity and oral hygiene measures is low among this group, leading to poor practice of oral hygiene measures, which outcomes to oral diseases. Implementation of health education program orphan children who are living in orphanages is important. the aim of this study is to evaluate the effectiveness of health education program on the knowledge and practice of orphan children. 80 children were enrolled in this study from different orphanages in Alexandria, Egypt. Knowledge and practice were evaluated before and after intervention using predesigned questionnaire, and oral hygiene was evaluated using simplified oral hygiene index

DETAILED DESCRIPTION:
Background: Dental caries is a lifetime disease, with highest priority risk group between 11-14 years of age group. Environmental factors such as culture, socioeconomic status, life style and dietary pattern can have a greater impact on caries-resistance or development. It has been well-documented in dentistry and other health areas that correct health information or knowledge alone does not necessarily lead to desirable health behaviors. However knowledge gained may serve as a tool to empower population groups with accurate information about health and health care technologies, enabling them to take action to protect their health. According to global review of oral health, despite great improvements in the oral health of populations in several countries, the oral problem persists. This is particularly among underprivileged groups, in both developed and developing countries. One of the known high-risk groups is orphans. An orphan is defined as a child under 18 years, who has lost his father, mother, or both In developing countries like Egypt, there is little access to oral healthcare due to a lack of knowledge, insufficient financial resources, and inadequate dental manpower in the national healthcare system Aim of the study: is to evaluate the effectiveness of oral health education programs on knowledge and practice of participated orphan children Materials and Methods: A specially designed questionnaire was used to assess the dental problems and existing oral hygiene maintenance practice among children between 6 - 12 years of age (n=80) in orphanages. DMFT [Decayed Missing Filled Teeth index (for permanent teeth)] and dft [ decayed filled teeth index ( for primary teeth) ], pre- and post-interventional intra-oral examinations was carried out to check their oral hygiene status which included and OHIS (Simplified Oral Hygiene Index).

Information regarding tooth cleaning habits was obtained by a questionnaire to the children themselves, before, immediately and after 6 months.

Statistical analysis Collected data will be analyzed using SPSS software

ELIGIBILITY:
Inclusion Criteria:

* Orphan children aged between 6-12 years old

Exclusion Criteria:

* children suffering from any systemic diseases acute or chronic, congenital abnormalities, psychological or behavioral problems, or receiving medications

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Knowledge will be assessed using predesigned questionnaire | Knowledge was measured immediately and after 6 months
  The questionnaire consisted of 8 questions to collect data about the children knowledge about teeth number in each dentition, the parts of teeth and its function, causes of oral disease, and how to prevent it.

SECONDARY OUTCOMES:
Practice will be assessed using predesigned questionnaire | Practice was evaluated after 6 months
  practices were measured using a predesigned questionnaire, consisting of 6 questions to collected data about the children's practices regarding tooth brushing, flossing and eating habits.
oral hygiene | oral hygiene was evaluated after 6 months
  Oral hygiene was evaluated using the simplified oral hygiene index - scores were ranged from 0-6 and 6 is the poorest oral hygiene score

CONTACTS AND LOCATIONS:
Overall Officials: Inas M Karawia, Principal Investigator — Pharos University in Alexandria
Locations (1):
- Pharos University in Alexandria, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No